CLINICAL TRIAL: NCT06783608
Title: The Effect of Laughter Yoga on Postprandial Blood Glucose Levels, Disease Perception and Perceived Stress Level in Patients With Type 2 Diabetes Mellitus: Randomized Controlled Trial
Brief Title: Laughter Yoga on Blood Glucose Levels, Disease Perception and Perceived Stress Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hakime Aslan, Principal investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Abdurrahman Akçin
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Blood Glucose; Diabetes Mellitus; Laughter Yoga; Nursing; Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter yoga group (Experimental): Laughter yoga
  Interventions: Behavioral: Laughter yoga
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Laughter yoga — Laughter yoga was applied to the experimental group for 4 weeks, 2 days a week, for 8 sessions (each session duration is 30-45 minutes on average). Patients were asked to measure and record their blood glucose value before breakfast. The yoga session was started 30 minutes after breakfast, and after the session was completed, they were asked to measure and record their blood glucose value again at 120 minutes after breakfast.
  Arms: Laughter yoga group

SUMMARY:
Aim This study was conducted to evaluate the effect of laughter yoga on blood glucose level, disease perception and perceived stress level in patients with Type 2 diabetes mellitus.

Method The study was conducted using a randomized controlled experimental design with a pre-test and post-test. The population of the study was followed up with the diagnosis of Type 2 diabetes mellitus (T2DM) in the endocrine outpatient clinics of a hospital in the western region of Turkey. The sample consisted of 100 patients (laughter yoga group=50, control group=50) determined by power analysis. Participants were assigned to each group through a process of simple randomization. Data collection was facilitated using a "Patient Identification Form,", "The Brief Disease Perception Scale," and " The Perceived Stress Scale".

DETAILED DESCRIPTION:
During the research process, in the laughter yoga group participated in eight laughter yoga sessions. while the patients in the control group continued to receive routine care practices.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2DM for at least 6 months,
* Able to use computer and/or mobile applications,
* At least primary education graduate,
* Using oral antidiabetic drugs,
* No diagnosed psychiatric illness,
* No communication problems,
* Patients who volunteered to participate in the study were included.

Exclusion Criteria:

* Using Parenteral Insulin,
* The one who doesn't attend all the yoga sessions,
* Patients with physical conditions that prevent them from participating in laughter yoga sessions (respiratory distress, persistent cough, veritgo, severe heart disease, hemeroid, hernia of any kind, severe back pain, urinary incontinence, epilepsy, bleeding tendency, thrombocytopenia and deformity visible on examination),
* Patients taking medication or other nonpharmacological methods to reduce stress,
* Patients who did not want to participate in the study were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
The effect of Laghter yoga on blood glucose value | 1 month
  Blood glucose follow-up charts were given to the patients and they were informed about the measurement times. In this study, the blood glucose measurement of the patients was before breakfast and after the sessions (after breakfast in the control group). Postprandial blood glucose (2-hour postprandial) was performed twice. Measurements were measured from fingertips by enzyme colorimetric assay using a blood glucose meter by the individuals themselves.
  Patients were asked to measure and record their blood glucose level before breakfast. The yoga session was started 30 minutes after breakfast, and after the session was completed, they were asked to measure and record their blood glucose level again at 120 minutes after breakfast.

SECONDARY OUTCOMES:
The effect of Laghter yoga on disease perception | 1 month
  'The Brief Disease Perception Scale (B-IPQ)' was used to evaluate how diabetic patients perceive the disease. During the data collection process, the scale was applied to the patients in both groups and pre-test data were collected. One month later, the scale was applied again and the change in disease perceptions was evaluated.
  The Brief Disease Perception Scale (B-IPQ) The Brief Illness Perception Questionnaire (B-IPQ), developed by Broadbent and colleagues, examines how individuals perceive their illness. It comprises nine items. Each item investigates a different aspect of illness perception. Respondents are asked to rate each item on a scale from 0 to 10. The Turkish version of the B-IPQ was validated and deemed reliable by Karataş and others in 2017.Scores between 0 and 80 can be obtained from the scale. As the disease perception score increases, the level of being affected by the disease and the level of seeing the disease as worrying also increases.

OTHER OUTCOMES:
The effect of Laghter yoga on percived stress | 1 month
  The Perceived Stress Scale (PSS) was used to evaluate the stress perceived by diabetic patients. During the data collection process, the scale was applied to patients in both groups and pre-test data were collected. One month later, the scale was applied again and the change in perceived stress was evaluated.
  The Perceived Stress Scale (PSS) The Perceived Stress Scale (PSS) was developed by Cohen, Kamarck, and Mermelstein. The Turkish validation and reliability of the scale was conducted by Eskin and colleagues. This tool includes 14 questions that assess individuals' perception of stress in various scenarios in their life. Using a five-point Likert scale, responses range from 0 (never) to 4 (very often). Scores between 0-56 can be obtained from the scale. There is no cut-off point in the scale, and an increase in the score indicates that the stress perception of the individual is high.

CONTACTS AND LOCATIONS:
Overall Officials: Hakime Aslan, Study Director — Inonu University
Locations (1):
- Hakime Aslan, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aslan H, Erci B. The effect of playing games with toys made with medical materials in children with cancer on pain during intravenous treatment. Palliat Support Care. 2022 Feb;20(1):84-93. doi: 10.1017/S1478951521000390. PMID 33947501